CLINICAL TRIAL: NCT04575467
Title: A 2-Stage Adaptive Design, Phase 2 Study to Evaluate the Efficacy, Safety and Tolerability of CBL-514 Injection for Reducing Abdominal and Thigh Subcutaneous Fat (Stage 1)
Brief Title: A Study to Evaluate the Efficacy, Safety and Tolerability of CBL-514 Injection for Reducing Subcutaneous Fat (Stage 1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Caliway Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CBL-0202
Record Dates: First submitted 2020-08-19; First posted 2020-10-05 (Actual); Results first posted 2024-03-28 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Subcutaneous Fat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CBL-514 320 mg (Experimental): CBL-514 will be administered via injection into the thigh subcutaneous adipose layer.
  Interventions: Drug: CBL-514
- CBL-514 480 mg (Experimental): CBL-514 will be administered via injection into the abdomen subcutaneous adipose layer.
  Interventions: Drug: CBL-514
- CBL-514 640 mg (Experimental): CBL-514 will be administered via injection into the abdomen subcutaneous adipose layer.
  Interventions: Drug: CBL-514
- CBL-514 800 mg (Experimental): CBL-514 will be administered via injection into the abdomen subcutaneous adipose layer.
  Interventions: Drug: CBL-514

INTERVENTIONS:
Drug: CBL-514 — CBL-514 will be administered via injection into the subcutaneous adipose layer.

SUMMARY:
The Stage 1 of this phase 2 study is an open-label single ascending dose (SAD) study. The primary objectives are to evaluate the safety and tolerability of injection lipolysis with CBL-514. It will be followed by a parallel-arm multiple-dose design in Stage 2.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) >18.5 and <32 kg/m2 and body weight ≥50 kg at Screening and Day 1.
2. Subject has sufficient thigh subcutaneous fat thickness of at least 1.50 cm (15.0 mm) and up to 5.00 cm (50.0 mm) measured by ultrasound, surrounding the center of treatment area at Screening and Day 1.
3. Subject has stable body weight (identified as ≤ 5% weight change) for at least 3 months before Screening and during the study.
4. Subject who has maintained a stable lifestyle (e.g. exercise, eating patterns, and smoking habit) for at least 3 months before Screening and during the study.
5. Voluntarily signs the Informed Consent Form (ICF) and, in the opinion of the Investigator or delegate, is physically and mentally capable of participating in the study, and willing to adhere to study procedures.

Exclusion Criteria:

1. Female subject of childbearing potential who is not willing to commit to an acceptable contraceptive regimen with her partner from the time of Screening and throughout study participation until 90 days after the last investigational product (IP) dose, or who is currently pregnant or lactating. Male subject who is not willing to commit to an acceptable contraceptive method.

   Females who have been surgically sterilized (hysterectomy or bilateral oophorectomy) or who are post-menopausal (e.g., defined as at least 50 years with ≥12 months of amenorrhea with a follicle stimulating hormone (FSH) >40 IU/L) are considered to be of non-childbearing potential. Subjects who are not of childbearing potential are not required to use contraception.
2. Subject diagnosed with coagulation disorders or is receiving anticoagulant/antiplatelet therapy or medications or dietary supplements, which impede coagulation or platelet aggregation.
3. Subject has fasting hemoglobin A1c (HbA1c) ≥ 9%, delayed would healing, or any diabetic risks which, in the opinion of Investigator, is inappropriate to participate in the study.
4. Subject has a clinically significant cardiovascular disease and abnormal findings in electrocardiogram (ECG).
5. Subject with active or prior history of malignancies within 5 years before Screening or being worked-up for a possible malignancy. Except adequately treated basal cell carcinoma of skin and in situ squamous cell carcinoma of skin would be eligible as per Investigator's discretion.
6. Subject with a history of human immunodeficiency virus (HIV)-1, infection or subjects with active HIV infection at Screening with positive HIV antigen/antibody (Ag/Ab) combo test.
7. Subjects with any hepatic medical condition that would interfere with assessment of safety or efficacy or compromise the subject's ability to undergo study procedures or provide informed consent.
8. Subject has abnormal skin or local skin conditions at the treatment area, which in the opinion of Investigator, is inappropriate to participate in the study, including but not limited to any of the following:

   1. Skin manifestations of a systemic disease,
   2. Any abnormality of the skin or soft tissues of the area to be treated,
   3. Grade III cellulite (Nürnberger and Muller scale, Nürnberger F, 1978) at the area to be treated,
   4. Skin folding on treatment area when the subject is in the supine position,
   5. Sensory loss or dysesthesia in the area to be treated,
   6. Evidence of any cause of enlargement in the area to be treated other than localized subcutaneous fat,
   7. Tattoos on the area to be treated.
9. Subject who has undergone the following procedures:

   1. Previous surgery in the anticipated treatment area,
   2. Cardiac pacemakers or any implantable electrical device,
   3. Metal implants of any type in the area to be treated,
   4. Esthetic procedure i.e. liposuction to the region to be treated,
   5. Esthetic procedure e.g. cryolipolysis, ultrasonic lipolysis, low level laser therapy (LLLT), lipolysis injection to the region to be treated within 12 months before Screening or during the study.
10. Subject is on prescription or over-the-counter (OTC) weight reduction medication or weight reduction programs within 3 months before Screening or during the study.
11. Subject is undergoing chronic steroid or immunosuppressive therapy.
12. Requiring continual use of the following therapeutic agents during the study: S mephenytoin (Mesantoin), terfenadine (Teldane), buspirone (Buspar), fexofenadine (Fexotabs, Tefodine, Telfast, Xergic, Allegra, etc.).

    If a subject needs to use the above mentioned therapeutic agents during the study for any reason, these therapeutic agents should not be used at least for 48 hours prior to dosing and until 24 hours post-dose.
13. Unable to receive topical anesthesia (e.g., history of hypersensitivity to Benzocaine, lidocaine, or Tetracaine).
14. Subjects with known allergies or sensitivities to the IP or its components.
15. Subjects with inadequate liver function at Screening defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALKP), total bilirubin (TBIL), or gamma-glutamyl transferase (GGT) >3.0 × upper limit of normal (ULN).
16. Subjects with inadequate renal function, defined as abnormal serum creatinine, and urea >1.5 × ULN or estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2. Subjects who are currently on dialysis should be excluded.
17. Use of other investigational drug or device within 4 weeks prior to Screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Site, Melbourne, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CBL-514 320 mg | CBL-514 480 mg | CBL-514 640 mg | CBL-514 800 mg
Started | 6 | 7 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBL-514 320 mg | CBL-514 480 mg | CBL-514 640 mg | CBL-514 800 mg | Total
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 25
Age, Continuous [Median (Full Range); unit: years] | 52.5 [22 to 59] | 48 [19 to 56] | 31.5 [21 to 59] | 51.5 [33 to 61] | 51 [19 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 6 | 3 | 20
  Male | 0 | 2 | 0 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 7 | 5 | 6 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 6 | 5 | 4 | 4 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 6 | 7 | 6 | 6 | 25
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 26.08 (1.95) | 25.16 (2.51) | 26.15 (3.74) | 25.97 (2.66) | 25.81 (2.64)
Weight [Mean (Standard Deviation); unit: kg] | 69.46 (7.58) | 75.25 (12.70) | 65.93 (9.01) | 75.48 (5.80) | 71.68 (9.65)

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events
Description: Number of treatment emergent adverse events (TEAEs)
Time Frame: Up to 4 weeks after treatment
Population: Safety Population
Measure: Number; unit: number of events
Arm/Group | CBL-514 320 mg | CBL-514 480 mg | CBL-514 640 mg | CBL-514 800 mg
Number analyzed (Participants) | 6 | 7 | 6 | 6
number of events | 103 | 57 | 69 | 61

2. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Values
Description: The clinical laboratory tests include Biochemistry, Hematology, Coagulation and Urinalysis test
Time Frame: Up to 4 weeks after treatment
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CBL-514 320 mg | CBL-514 480 mg | CBL-514 640 mg | CBL-514 800 mg
Number analyzed (Participants) | 6 | 7 | 6 | 6
Participants | 0 | 0 | 0 | 1

3. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital signs measurements include temperature, pulse rate, blood pressure, and respiratory rate
Time Frame: Up to 4 weeks after treatment
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CBL-514 320 mg | CBL-514 480 mg | CBL-514 640 mg | CBL-514 800 mg
Number analyzed (Participants) | 6 | 7 | 6 | 6
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG)
Description: ECG parameters include heart rate, RR interval, PR interval, QT interval, QTc interval, and QRS interval
Time Frame: Up to 4 weeks after treatment
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CBL-514 320 mg | CBL-514 480 mg | CBL-514 640 mg | CBL-514 800 mg
Number analyzed (Participants) | 6 | 7 | 6 | 6
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examination
Description: Physical examinations include assessment of cardiovascular, respiratory, gastrointestinal, and neurological systems
Time Frame: Up to 4 weeks after treatment
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | CBL-514 320 mg | CBL-514 480 mg | CBL-514 640 mg | CBL-514 800 mg
Number analyzed (Participants) | 6 | 7 | 6 | 6
Participants | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Injection Site Reactions
Description: Injection site reactions include but not limited to redness, swelling, bruising, tenderness, itching, pain, warmth, discoloration and hardness
Time Frame: Up to 4 weeks after treatment
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CBL-514 320 mg | CBL-514 480 mg | CBL-514 640 mg | CBL-514 800 mg
Number analyzed (Participants) | 6 | 7 | 6 | 6
Participants | 6 | 7 | 6 | 6

7. Secondary Outcome: Change in Subcutaneous Fat Thickness
Description: Change in subcutaneous fat thickness as measured by ultrasound compared to Baseline. No efficacy assessments were done for Group 1 of Stage 1 study.
Time Frame: Up to 4 weeks after treatment
Population: ITT Population (Data not collected for participants that received the 320 mg injection)
Measure: Mean (Standard Deviation); unit: Absolute Change (mm) from Baseline
Arm/Group | CBL-514 480 mg | CBL-514 640 mg | CBL-514 800 mg
Number analyzed (Participants) | 7 | 6 | 6
Absolute Change (mm) from Baseline | -4.77 (2.29) | -4.85 (2.02) | -2.98 (2.83)
Statistical Analysis 1: Comparison: CBL-514 480 mg; Test type: Superiority; p < 0.01, Paired t-test; Mean absolute fat thickness difference = -4.77, 95% CI 2-sided [-7.17 to -2.37], Standard Deviation 2.29
Statistical Analysis 2: Comparison: CBL-514 640 mg; Test type: Superiority; p < 0.01, Paired t-test; Mean absolute fat thickness difference = -4.85, 95% CI 2-sided [-6.97 to -2.73], Standard Deviation 2.02
Statistical Analysis 3: Comparison: CBL-514 800 mg; Test type: Superiority; p < 0.05, Paired t-test; Mean absolute fat thickness difference = -2.98, 95% CI 2-sided [-5.95 to -0.01], Standard Deviation 2.83

8. Secondary Outcome: Change in Subcutaneous Fat Volume
Description: Change in subcutaneous fat volume over the treated area as measured by ultrasound compared to Baseline. No efficacy assessments were done for Group 1 of Stage 1 study.
Time Frame: Up to 4 weeks after treatment
Population: ITT Population (Data not collected for participants that received the 320 mg injection)
Measure: Mean (Standard Deviation); unit: Absolute change (mL) from Baseline
Arm/Group | CBL-514 480 mg | CBL-514 640 mg | CBL-514 800 mg
Number analyzed (Participants) | 7 | 6 | 6
Absolute change (mL) from Baseline | -114.40 (54.88) | -155.20 (64.70) | -119.17 (113.11)
Statistical Analysis 1: Comparison: CBL-514 480 mg; Test type: Superiority; p < 0.01, Paired t-test; Mean absolute fat volume difference = -114.40, 95% CI 2-sided [-171.99 to -56.81], Standard Deviation 54.88
Statistical Analysis 2: Comparison: CBL-514 640 mg; Test type: Superiority; p < 0.01, Paired t-test; Mean absolute fat volume difference = -155.20, 95% CI 2-sided [-223.10 to -87.30], Standard Deviation 64.70
Statistical Analysis 3: Comparison: CBL-514 800 mg; Test type: Superiority; p < 0.05, Paired t-test; Mean absolute fat volume difference = -119.17, 95% CI 2-sided [-237.86 to -0.47], Standard Deviation 113.11

ADVERSE EVENTS:
Time Frame: Up to 4 weeks after treatment
Arm/Group | CBL-514 320 mg | CBL-514 480 mg | CBL-514 640 mg | CBL-514 800 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBL-514 320 mg (N=6) | CBL-514 480 mg (N=7) | CBL-514 640 mg (N=6) | CBL-514 800 mg (N=6)
Closed head injury with post concussive symptoms (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBL-514 320 mg (N=6) | CBL-514 480 mg (N=7) | CBL-514 640 mg (N=6) | CBL-514 800 mg (N=6)
Injection site erythema (General disorders) | 6 (12) | 7 (7) | 6 (6) | 6 (6)
Injection site bruising (General disorders) | 6 (12) | 6 (6) | 6 (6) | 6 (8)
Injection site pain (General disorders) | 6 (18) | 6 (11) | 6 (13) | 6 (13)
Injection site swelling (General disorders) | 6 (12) | 6 (6) | 6 (6) | 6 (6)
Injection site pruritus (General disorders) | 4 (10) | 7 (7) | 6 (6) | 6 (7)
Injection site warmth (General disorders) | 6 (12) | 5 (5) | 3 (3) | 6 (6)
Injection site discolouration (General disorders) | 6 (12) | 6 (6) | 3 (3) | 1 (1)
Injection site induration (General disorders) | 6 (13) | 4 (4) | 2 (3) | 4 (5)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 1 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT04575467/Prot_002.pdf
  • Statistical Analysis Plan (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT04575467/SAP_003.pdf